CLINICAL TRIAL: NCT01221220
Title: Environmental Strategies & Behavior Change to Reduce Overeating in Obese Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Thomas Robinson, Irving Schulman, MD Endowed Professor in Child Health; Professor of Pediatrics and of Medicine and CHP/PCOR Associate, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SU-08302010-6809; R01HL096015 (NIH)
Record Dates: First submitted 2010-10-13; First posted 2010-10-14 (Estimated); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Behavioral Treatment (Active Comparator): Six-month, family-based, group, behavioral weight control program
  Interventions: Behavioral: Standard Packard Pediatric Weight Control Program
- Behavioral Treatment plus Environmental Strategies (Experimental): Six-month, family-based, group, behavioral weight control program plus home-based environmental intervention
  Interventions: Behavioral: Standard Packard Pediatric Weight Control Program plus Home-based advising on environmental changes

INTERVENTIONS:
Behavioral: Standard Packard Pediatric Weight Control Program — Six-month, family-based, group, behavioral weight control program
  Arms: Behavioral Treatment
Behavioral: Standard Packard Pediatric Weight Control Program plus Home-based advising on environmental changes — Six-month, family-based, group, behavioral weight control program plus Home-based Environmental strategies intervention
  Arms: Behavioral Treatment plus Environmental Strategies

SUMMARY:
There is a need for effective weight control methods for obese children. Environmental strategies such as reducing the size of dishware and serving utensils, storing food out of view and reducing food consumption while watching television may reduce food intake without requiring conscious, cognitive self-control. The investigators propose to test these methods when added to a current state-of-the-art behavioral program.

DETAILED DESCRIPTION:
Single blind study with outcome assessors (data collectors)and investigators masked (blinded) to intervention assignment. Analysis is intention-to-treat.

ELIGIBILITY:
Inclusion Criteria:Inclusion criteria: 8-15 year old obese children (BMI ≥ 95th percentile on the 2000 CDC BMI reference) on the date of randomization. Our standard Stanford Pediatric Weight Control Program eligibility criteria will apply: both child and parent/guardian must want to join, both child and at least one parent/guardian must agree to attend sessions, and must agree to not miss more than 2 consecutive sessions. As we interested in testing generalizable strategies for weight control in diverse populations, the eligibility criteria are designed to be liberal, to maximize the generalizability of the results, but also maintain the internal validity of the test of the intervention. Exclusion Criteria:Exclusions: To enhance internal validity, children will not be eligible if they:

1. have been diagnosed with a medical condition affecting growth (a genetic or metabolic disease/syndrome associated obesity, Type 1 diabetes, Type 2 diabetes taking medication, chronic gastrointestinal diseases, Chronic renal diseases, uncorrected structural heart disease, heart failure, heart transplant, anorexia nervosa or bulimia nervosa or binge eating disorder [present or past], AIDS or HIV infection, pregnancy);
2. are taking medications affecting growth (systemic corticosteroids more than 2 weeks in the past year, insulin, oral hypoglycemics, thyroid hormone, growth hormone);
3. have a condition limiting their participation in the interventions (e.g., unable to participate in routine physical education classes at school, requiring oxygen supplementation for exertion, developmental or physical disability preventing participation in interventions, children or parents/guardians who cannot medically participate in mild dietary restrictions and/or increased physical activity for any reason);
4. have a condition limiting participation in the assessments (child or primary caregiver not able to read surveys in English or Spanish, child two or more grade levels delayed in school for reading and writing in his/her native language);
5. are unable to read, understand or complete informed consent in English or Spanish;
6. plan to move from the San Francisco Bay Area within the next 18 months.

Ages: 8 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 174 (Actual)
Dates: Start 2010-09; Primary Completion 2014-10-15 (Actual); Study Completion 2014-10-15 (Actual)

PRIMARY OUTCOMES:
Body Mass Index (BMI) | 18 months post randomization

SECONDARY OUTCOMES:
Waist Circumference | 6 months and 18 months post randomization
Triceps skinfold | 6 months and 18 months post randomization
Resting heart rate | 6 months and 18 months post randomization
Dietary intake/ meals eaten with television | 6 months and 18 months post randomization
Weight concerns | 6 months and 18 months post randomization
Depressive symptoms | 6 months and 18 months post randomization
Daily energy intake | 6 months and 18 months post randomization
Physical Activity | 6 months and 18 months post randomization
Systolic and diastolic blood pressure | 6 months and 18 months post randomization
Fasting blood lipids, insulin/glucose metabolism | 6 months and 18 months post randomization
Body Mass Index (BMI) | 6 months post randomization

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Robinson, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States